CLINICAL TRIAL: NCT06094153
Title: Randomized Controlled Trial on Prebiotic Effects on Gut Microbiota, Gut Comfort and Immune Function
Brief Title: Prebiotic Effects on Gut Microbiota, Gut Comfort and Immune Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyowa Hakko Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-005
Record Dates: First submitted 2023-07-11; First posted 2023-10-23 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Gastrointestinal Diseases
Keywords: Prebiotics
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- HMO 1 (Experimental)
  Interventions: Dietary Supplement: HMO 1
- HMO 2 (Experimental)
  Interventions: Dietary Supplement: HMO 2

INTERVENTIONS:
Dietary Supplement: Placebo — Consume placebo (Maltodextrin) once daily before going to bed for 28 days
  Arms: Placebo
Dietary Supplement: HMO 1 — Consume HMO 1 (Dietary supplement) once daily before going to bed for 28 days
  Arms: HMO 1
Dietary Supplement: HMO 2 — Consume HMO 2 (Dietary supplement) once daily before going to bed for 28 days
  Arms: HMO 2

SUMMARY:
Human Milk Oligosaccharides (HMOs) are the third most abundant class of nutrients in human milk. Studies investigating the effects of dietary HMOs in infants have shown various health and developmental benefits such as the development of the early gut microbiome (by favouring colonisation of beneficial Bifidobacterium, Lactobacillus, and Bacteroides), the development of the immune system, general infant growth, protection against infectious diseases and allergies, and stimulation of cognitive development. Only a limited number of studies have been conducted in adults, showing intake of HMOs stimulates the growth of gut Bifidobacterium in healthy adults.

DETAILED DESCRIPTION:
The current study aims to investigate the effects of a 4-week intervention with two HMOs on gut microbiome composition, immune function and gastrointestinal symptoms in healthy adults with mild to moderate gastrointestinal complaints. The study will be conducted as a partially decentralized, double-blind, randomized, placebo-controlled, parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 and ≤ 55 years
* Male/female
* Total score of >2 on the Gastrointestinal Symptom Rating Scale (GSRS)
* Body Mass Index 18-30 kg/m2
* Stable body weight (± 5%) for at least 6 months
* Stable lifestyle and dietary habits within the 4 weeks prior and during study period
* Owns device (computer, smartphone, tablet) with access to the internet
* Adequate fluency in the English language to understand the inform consent process, study instructions and study assessments
* Sufficient vision and hearing to complete study procedures
* Willing and able to participate, follow the study procedures and to give written informed consent

Exclusion Criteria:

* History (< 6 months prior to the study) or presence of severe gastrointestinal, metabolic, immunological, psychiatric disorder, or major surgery
* Current or past (< 4 weeks) use of prescription, over-the-counter, or traditional medication, or dietary supplements with a relevant impact on GI system or on visceral motility
* Having received antibiotic treatment < 4 weeks prior to study
* Alcohol intake >1 units/day
* Currently pregnant or pregnancy in past 6 months
* Use of pro/prebiotics < 4 weeks prior to study start
* Fully vegetarian/vegan diet < 4 weeks prior to study start
* High habitual vegetable and fruit intake (> 2 servings of fruits and >2 servings of vegetables per day) < 4 weeks prior to study start
* Lactose intolerance
* Maltodextrin allergy
* Members of the research team or their immediate family members. Immediate family member is defined as spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Relative abundance of Bifidobacterium in the gut | 4 weeks

SECONDARY OUTCOMES:
Relative abundance of other bacterial taxa in the gut | 4 weeks
Gut microbiome functional potential (functional metagenomics analyses) | 4 weeks
Stool Human Milk Oligossacharides level | 4 weeks
Concentration of immune parameters panel in blood (OLINK Target 96 Inflammation panel) | 4 weeks

OTHER OUTCOMES:
Gastrointestinal Symptoms Questionnaire | 4 weeks
Depression Anxiety Stress Scale (DASS)-21 items | 4 weeks
Digestion-associated Quality of Life Questionnaire (DQLQ) | 4 weeks
Bristol stool chart | 4 weeks
  Stool consistency ranging from Type 1 to Type 7
Clinical chemistry and haematology analyses for safety analysis | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Institute for Clinical Trials, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprenger N, Tytgat HLP, Binia A, Austin S, Singhal A. Biology of human milk oligosaccharides: From basic science to clinical evidence. J Hum Nutr Diet. 2022 Apr;35(2):280-299. doi: 10.1111/jhn.12990. Epub 2022 Feb 2. PMID 35040200
- [Background] Elison E, Vigsnaes LK, Rindom Krogsgaard L, Rasmussen J, Sorensen N, McConnell B, Hennet T, Sommer MO, Bytzer P. Oral supplementation of healthy adults with 2'-O-fucosyllactose and lacto-N-neotetraose is well tolerated and shifts the intestinal microbiota. Br J Nutr. 2016 Oct;116(8):1356-1368. doi: 10.1017/S0007114516003354. Epub 2016 Oct 10. PMID 27719686